CLINICAL TRIAL: NCT05864378
Title: The Impact of Point-of-care Ultrasound on the Diagnosis and Management of Small Bowel Obstruction in the Emergency Department: a Retrospective Observational Single-center Study
Brief Title: POCUS for Small Bowel Obstruction in the ED: a Retrospective Study
Acronym: SBOCUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Carmine Cristiano Di Gioia, Attending physician, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: SBOCUS2023
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Small Bowel Obstruction; Point of Care Ultrasound
Keywords: POCUS; SBO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The POCUS group: Patients who were evaluated by ED physicians who perform POCUS intestinal loops examination as part of their clinical practice
- The non-POCUS group: Patients who were evaluated by ED physicians who do not perform POCUS intestinal loops examination for any reason

SUMMARY:
This study protocol aims to evaluate the impact of point-of-care ultrasound (POCUS) on the diagnosis and management of small bowel obstruction (SBO) in the emergency department (ED). SBO is a potentially life-threatening condition that requires prompt diagnosis and management. Currently, the diagnosis of SBO is based on clinical evaluation and imaging tests, including plain abdominal radiography and computed tomography (CT) scan. POCUS is a bedside imaging technique that is rapid, non-invasive, repeatable, cost-effective and radiation-free, and can provide valuable information for the diagnosis and management of SBO. The primary objective of this study is to compare the time to diagnosis of SBO between patients who undergo POCUS intestinal loops examination and those who do not undergo POCUS in the ED. The secondary objectives include comparing the hospital length of stay, the rate of surgical intervention, the rate of complications, and the mortality rate between the two groups. This is a monocentric retrospective cohort study that will include all adult patients (> 18 years old) who presented to the ED with suspected SBO. The study population will be divided into two groups: the POCUS group and the non-POCUS group. The sample size calculation will be based on the assumption of a 30% reduction in the time to diagnosis of SBO in the POCUS group compared to the non-POCUS group, with a power of 80%. The results of this study may provide more robust evidence on the diagnostic accuracy and impact of POCUS for SBO in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Clinical suspicion of SBO based on history and physical examination
* Plain abdominal radiography (AXR) or CT scan performed in the ED

Exclusion Criteria:

* Pregnancy
* Known bowel obstruction
* Previous abdominal surgery within 30 days
* Refusal or inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be divided into two groups:
  1. The POCUS group: patients who were evaluated by ED physicians who perform POCUS intestinal loops examination as part of their clinical practice
  2. The non-POCUS group: patients who were evaluated by ED physicians who do not perform POCUS intestinal loops examination for any reason.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis of SBO by POCUS or CT scan | All patients will be seen by the emergency physician within 6 hours of admission to the emergency department.
  The primary outcome will be the time to diagnosis of SBO by POCUS or CT scan, defined as the interval between the ED arrival and the confirmation of SBO by either imaging modality, comparing the two groups.

SECONDARY OUTCOMES:
The hospital length of stay | Patients will be followed up for a maximum of 2 months from admission to the emergency department, until discharge or death.
  The interval between the ED arrival and the hospital discharge
The rate of surgical intervention | Patients will be followed up for a maximum of 2 months from admission to the emergency department, until discharge or death.
  The proportion of patients who underwent laparotomy or laparoscopy for SBO
The rate of complications | Patients will be followed up for a maximum of 2 months from admission to the emergency department, until discharge or death.
  The proportion of patients who developed bowel ischemia, perforation, peritonitis or sepsis during their hospitalization
The mortality rate | Patients will be followed up for a maximum of 2 months from admission to the emergency department, until discharge or death.
  The proportion of patients who died during their hospitalization or within 30 days after their ED arrival